CLINICAL TRIAL: NCT03617055
Title: Early Predictor of Acute Kidney Injury in Newborns With Perinatal Asphyxia
Brief Title: Acute Kidney Injury in Newborns With Perinatal Asphyxia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, M. A. Sabra, Mohammed Abdel tawab sabra, Assiut University
Other Study IDs: AKIPA
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Acute Kidney Injury
Keywords: kidney injury, asphyxia,cystatin c
MeSH Terms: conditions — Acute Kidney Injury; Asphyxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum cystatin c — Blood sample for serum cystatin c will be taken on the first and third days of life for all neonates with clinical or laboratory signs of perinatal asphyxia who are admitted to NICU for early detection of AKI in the study group.

SUMMARY:
The aim of the study is to investigate the role of serum cystatin C (sCysC) as an early predictor for both diagnosis and short term outcome evaluation of acute kidney injury (AKI) in neonates with perinatal asphyxia admitted to Neonatal Intensive Care Unit (NICU) of Assiut University Children Hospital

DETAILED DESCRIPTION:
Acute Kidney Injury is defined as the inability of the kidneys to excrete nitrogenous waste products and maintain fluid and electrolyte homeostasis. It is fairly common in newborn population and is a major contributor factor of neonatal mortality and morbidity.

The most common form of Acute Kidney Injury in neonates is prerenal failure due to renal hypo-perfusion or ischemia. Pre-renal failure may result in intrinsic kidney failure if it is not treated promptly. The kidneys of neonates are particularly susceptible to hypo-perfusion because of the physiologic characteristics of neonatal kidneys, including high renal vascular resistance, high plasma renin activity, low glomerular filtration, decreased intra-cortical perfusion rate and decreased reabsorption of sodium in the proximal tubules in the first days of a neonatal life. Thus, newborn infants are vulnerable to acute tubular necrosis or cortical necrosis.

The cause of Acute Kidney Injury in neonates is of multi-factorial etiology and, usually, there is one or more associated contributing factor. In most studies, perinatal asphyxia and sepsis are the most commonly associated conditions.

Perinatal asphyxia is defined as abnormal neurological incident resulting in neonatal hypoxic ischemic encephalopathy , which occurs usually due to brain hypoxia and ischemic incidents. Perinatal asphyxia can result in multi-organ dysfunction through redirection of cardiac output to maintain cerebral, cardiac, and adrenal perfusion while potentially compromising perfusion to non-vital organs including kidneys, this causing Acute Kidney Injury.

The incidence of Acute Kidney Injury after Perinatal asphyxia in term neonates was shown to be around 30% to 56%. Early detection of Acute Kidney Injury could optimize and improve patient outcomes. therefore, the use of biomarkers to predict renal damage has been of interest. Serum creatinine is the most commonly used clinical measure of renal function; however, it is a poor diagnostic marker and its utility is further questionable in neonates since kidneys undergo maturational changes in postnatal period.

Human Cystatin C is a low molecular weight protein, belonging to the cystatin superfamily of protease inhibitors, which is produced at a constant rate in all nucleated cells. Cystatin C is freely filtered through the glomerular membrane, then completely reabsorbed and degraded by the proximal tubule. Serum Cystatin C is being promoted as a more accurate estimate of neonatal glomerular filtration rate.

Acute Kidney Injury was diagnosed on the basis of changes in the serum creatinine level according to the modified neonatal Acute Kidney Injury of Kidney Disease Improving Global Outcome definition (Table 1). AKI was defined as an increase in the serum creatinine level by ≥ 0.3 mg/dL within 48 hours or ≥ 1.5 times from the baseline within 7 days.

Newborns are unique in that the serum creatinine level immediately after birth often reflects maternal levels. Studies have reported that the mean serum creatinine level in preterm infants rises during the first two days of postnatal life, reaches a plateau for a few days, and then decreases thereafter .Therefore, the baseline serum creatinine level was defined as the lowest previous serum creatinine level after 24 hours of age.

TABLE 1 Acute Kidney Injury of Kidney Disease Improving Global Outcome definition:

Stage serum creatinine Urine Output 0 No change or rise < 0.3 mg/dL. ≥ 0.5 mL/kg/h.

1. rise ≥ 0.3 mg/dL within 48 h or rise ≥1.5-1.9 × reference level* within 7 days. < 0.5 mL/kg/h for 6 to 12 h.
2. rise ≥ 2.0-2.9 × reference level * < 0.5 mL/kg/h for ≥ 12 h.
3. rise ≥ 3 × reference level * or serum creatinine level ≥ 2.5 mg/dL or Receipt of dialysis. < 0.3 mL/kg/h for ≥ 24 h or anuria for ≥ 12 h.

   * Reference level will be defined as the lowest previous serum creatinine.

The goal of Acute Kidney Injury management in newborns is to maintain homeostasis until the renal functions return, and is accomplished by addressing fluid and electrolyte imbalance, nutritional needs, and acidosis.Unfortunately, available data on the long-term outcome of neonatal Acute Kidney Injury patients is limited.

The short-term outcome of therapy for Acute Kidney Injury in newborns is dependent on the underlying etiology of Acute Kidney Injury, the involvement of other organs and the availability of renal replacement therapy. As expected, mortality is more frequent and morbidity is much worse in neonates with multi-organ failure.

ELIGIBILITY:
Inclusion Criteria:

* all full term neonates who are admitted to neonatal intensive care unit of Assiut University Children Hospital through the period from Jan. 2019 to Jan. 2020 with documented perinatal asphyxia

Exclusion Criteria:

preterm neonates < 37 weeks, neonates who died within the first 24 hours of admission, neonates with any congenital anomalies like skeletal, renal or urinary tract, neonates with AKI for any cause other than asphyxia and neonates with maternal history of renal failure .

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all full term neonates with documented perinatal asphyxiaby by one of the following indicators: (i) Presence of a sentinel hypoxic event immediately before or during delivery; (ii) History of fetal distress (bradycardia, late decelerations, absence of heart rate variability); (iii) Need for neonatal resuscitation at delivery; (iv) 1-min Apgar score <3 or 5-min Apgar score <7; or metabolic acidosis (BE > 10 in cord blood).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
serum cystatin C (sCysC) as an early predictor of acute kidney injury (AKI) in neonates with perinatal asphyxia. | one year
  measuring serum cystatin c in neonates with perinatal asphyxia

SECONDARY OUTCOMES:
is to determine the incidence of Acute kidney injury in neonates with perinatal asphyxia. | one year

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdulkader RC, Liborio AB, Malheiros DM. Histological features of acute tubular necrosis in native kidneys and long-term renal function. Ren Fail. 2008;30(7):667-73. doi: 10.1080/08860220802212460. PMID 18704814
- [Background] Coca SG, Singanamala S, Parikh CR. Chronic kidney disease after acute kidney injury: a systematic review and meta-analysis. Kidney Int. 2012 Mar;81(5):442-8. doi: 10.1038/ki.2011.379. Epub 2011 Nov 23. PMID 22113526
- [Background] Mathur NB, Agarwal HS, Maria A. Acute renal failure in neonatal sepsis. Indian J Pediatr. 2006 Jun;73(6):499-502. doi: 10.1007/BF02759894. PMID 16816511
- [Background] Cuzzolin L, Fanos V, Pinna B, di Marzio M, Perin M, Tramontozzi P, Tonetto P, Cataldi L. Postnatal renal function in preterm newborns: a role of diseases, drugs and therapeutic interventions. Pediatr Nephrol. 2006 Jul;21(7):931-8. doi: 10.1007/s00467-006-0118-2. Epub 2006 May 25. PMID 16773403
- [Background] Subramanian S, Agarwal R, Deorari AK, Paul VK, Bagga A. Acute renal failure in neonates. Indian J Pediatr. 2008 Apr;75(4):385-91. doi: 10.1007/s12098-008-0043-4. Epub 2008 May 18. PMID 18536895
- [Background] Bona E, Hagberg H, Loberg EM, Bagenholm R, Thoresen M. Protective effects of moderate hypothermia after neonatal hypoxia-ischemia: short- and long-term outcome. Pediatr Res. 1998 Jun;43(6):738-45. doi: 10.1203/00006450-199806000-00005. PMID 9621982
- [Background] Oncel MY, Canpolat FE, Arayici S, Alyamac Dizdar E, Uras N, Oguz SS. Urinary markers of acute kidney injury in newborns with perinatal asphyxia (.). Ren Fail. 2016 Jul;38(6):882-8. doi: 10.3109/0886022X.2016.1165070. Epub 2016 Apr 7. PMID 27055689
- [Background] Durkan AM, Alexander RT. Acute kidney injury post neonatal asphyxia. J Pediatr. 2011 Feb;158(2 Suppl):e29-33. doi: 10.1016/j.jpeds.2010.11.010. PMID 21238703
- [Background] Bagshaw SM, Bellomo R. Early diagnosis of acute kidney injury. Curr Opin Crit Care. 2007 Dec;13(6):638-44. doi: 10.1097/MCC.0b013e3282f07570. PMID 17975383
- [Background] Kandasamy Y, Smith R, Wright IM. Measuring cystatin C to determine renal function in neonates. Pediatr Crit Care Med. 2013 Mar;14(3):318-22. doi: 10.1097/PCC.0b013e318271f4a5. PMID 23392363
- [Background] Jetton JG, Askenazi DJ. Acute kidney injury in the neonate. Clin Perinatol. 2014 Sep;41(3):487-502. doi: 10.1016/j.clp.2014.05.001. Epub 2014 Jul 22. PMID 25155722